CLINICAL TRIAL: NCT00590785
Title: Phase III Comparison of Adjuvant Chemotherapy W/High-Dose Cyclophosphamide Plus Doxorubicin (AC) vs Sequential Doxorubicin Fol by Cyclophosphamide (A-C) in High Risk Breast Cancer Patients With 0-3 Positive Nodes (Intergroup, CALGB 9394)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96-041; INT 0137; CALGB 9394
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: High Risk; Breast Cancer; Positive Nodes; Cyclophosphamide; Doxorubicin
Keywords: High Risk; Breast Cancer; Positive Nodes; Cyclophosphamide; Doxorubicin; 96-041
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Granulocyte Colony-Stimulating Factor; Filgrastim; Tamoxifen; Ciprofloxacin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: G-CSF; Drug: tamoxifen
- 2 (Experimental)
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: G-CSF; Drug: ciprofloxacin

INTERVENTIONS:
Drug: Doxorubicin — High-dose doxorubicin + cyclophosphamide (AC) x 6 cycles with G-CSF on Days 3 - 12 and followed in postmenopausal patients and hormone receptor-positive premenopausal patients by tamoxifen 20 mg daily for 5 years.
Drug: Cyclophosphamide — High-dose doxorubicin + cyclophosphamide (AC) x 6 cycles with G-CSF on Days 3 - 12 and followed in postmenopausal patients and hormone receptor-positive premenopausal patients by tamoxifen 20 mg daily for 5 years.
Drug: G-CSF — High-dose doxorubicin + cyclophosphamide (AC) x 6 cycles with G-CSF on Days 3 - 12 and followed in postmenopausal patients and hormone receptor-positive premenopausal patients by tamoxifen 20 mg daily for 5 years.
  Other Names: Filgrastim
Drug: tamoxifen — High-dose doxorubicin + cyclophosphamide (AC) x 6 cycles with G-CSF on Days 3 - 12 and followed in postmenopausal patients and hormone receptor-positive premenopausal patients by tamoxifen 20 mg daily for 5 years.
  Arms: 1
Drug: ciprofloxacin — High-dose sequential doxorubicin x 4 given with G-CSF on Days 3 - 12+ and followed by high-dose cyclophosphamide x 3 (A+C) given with G-CSF and ciprofloxacin on Days 3-12, followed in postmenopausal patients and hormone receptor-positive premenopausal patients by tamxifen 20 mg daily for 5 years.
  Arms: 2

SUMMARY:
To compare disease-free survival (DFS), overall survival (s), and toxicity of high-isk primary breast cancer patients with negative axillary lymph nodes or with one to three positive nodes treated with adjuvant high-dose chemotherapy with doxorubicin plus cyclophosphamide (AC), versus high-dose sequential chemotherapy with doxorubicin followed by cyclophosphamide (A-->C).

ELIGIBILITY:
* Patients must have been diagnosed with primary invasive adenocarcinoma of the breast. Those patients with the special types including pure tubular, mucinous and papillary carcinoma are not eligible. Patients must not have sarcoma, lymphoma, or apocrine, adenocystic or squamous cell cancer of the breast. Patients must not have recurrent invasive breast cancer. Metaplastic carcinomas are eligible as a variant form of adenocarcinoma.
* Patients must have undergone an axillary dissection, and at least 6 nodes must have een removed and examined. Nodal involvement by tumor must be negative or must not xceed three positive nodes.
* disease must be considered sufficiently high-risk by the investigator to justify the use of chemotherapy. To be eligible, disease must satisfy one of the following requirements:

  1. Tumor is both ER negative and PgR negative and greater than 1.0 cm in greatest diameter. Negative is defined as c 10 fmollmg cytosol protein if measured in these units; othennrise negative is defined according to institutional standards.
  2. Tumor that is greater than 2.0 cm in greatest diameter irrespective of hormone receptor status (including unknown).
  3. Tumor involves one to three axillary lymph nodes.
* Breast cancer was not locally advanced at diagnosis. This is left to investigator judgement, but generally should exclude patients with fixed tumors, fixed nodes, peau d'orange skin changes, skin ulcerations or inflammatory changes (T4 disease).
* Patient Is currently free of breast cancer (no evidence of disease). This is also left to investigator judgement, but generally should include no evidence of distant disease on chest x-ray or mgmmogram of the opposite breast prior to registration, within 3 months prior to surgery; and no gross or microscopically positive surgical margins noted in the final surgery or pathology reports. Patients with synchronous bilateral breast cancer may be considered, provided both breasts are treated with curative intent and that eligibility is based on the side with the most adverse prognostic features.
* Registration must be within 84 days of mastectomy, or within 84 days of axillary dissection if the patient's most extensive breast surgery was a breast sparing procedure. Patients not having mastectomy or breast sparing surgery are ineligible. Patients must not have had prior chemotherapy for this breast cancer. Patients must not have had systemic therapy of any type for a previous breast cancer.
* Patients must not have had external beam radiotherapy for this breast cancer prior to registration. Brachytherapy (interstitial radiation therapy) at the time of breast sparing procedure is acceptable and would not render the patient Ineligible. (If external beam radiotherapy is planned to be given with brachytherapy, it must be delayed until after chemotherapy is complete.) Patients whose most extensive breast surgery was a breast sparing procedure must be planning to receive radiotherapy after chemotherapy is complete.
* Patients must have adequate hematologic, hepatic, renal and cardiac function for high dose chemotherapy and adequate health for long-term follow-up. This must Include normal WBC (2 4,0001pl). neutrophll count (2 1,50O/pl), platelet count (2 Institutional lower limit of normal), and LVEF (left ventricular ejection fraction by institutional criteria); bilirubin within 1.5 times institutional upper limit of normal; creatinine within 1.5 times institutional upper limit of normal; and no serious disease other than breast cancer.
* Pregnant or nursing women may not participate. Men are ineligible. Women of childbearing potential must be planning to use effective contraception.
* All patients must be informed of the Investigational nature of this study and give written informed consent in accordance with institution and federal guidelines.
* At the time of registration, the date of institutional review board approval for this study must be provided to the Statistical Center.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1996-08-13; Primary Completion 1997-06-10 (Actual); Study Completion 2015-01-13 (Actual)

PRIMARY OUTCOMES:
To compare disease-free survival (DFS), overall survival (s), and toxicity of high-isk primary breast cancer patients with negative axillary lymph nodes or with one to three positive nodes. | Conclusion of the study

SECONDARY OUTCOMES:
To obtain tumor tissue for biologic studies. The details of these biologic studies will be described in a companion protocol or protocols to be developed through the Intergroup mechanism. | Conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Hudis, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org